CLINICAL TRIAL: NCT00169455
Title: A Phase IIIb, Partially Blind, Randomized, Placebo-controlled Study to Asses the Effect on Immunogenicity of Administration of Vaccine Without Buffering Agent and to Assess Heat Stability in Terms of Immunogenicity, Reactogenicity and Safety of GlaxoSmithKline Biologicals' Oral Live Attenuated Human Rotavirus (HRV) Vaccine Following a 0, 2 Month Schedule, in Healthy Infants Previously Uninfected With Human Rotavirus
Brief Title: Assess the Immunogenicity of the Human Rotavirus (HRV) Vaccine After Reconstitution Without Buffering Agent; & Evaluate the Immunogenicity, Reactogenicity & Safety of the Vaccine After Storage for 7 d at 37°C Following 2 Doses in Healthy Infants
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 103477
Record Dates: First submitted 2005-09-09; First posted 2005-09-15 (Estimated); Last update posted 2017-01-16 (Estimated); Status verified 2017-01

CONDITIONS: Rotavirus Gastroenteritis

INTERVENTIONS:
Biological: Live attenuated human rotavirus vaccine

SUMMARY:
Rotavirus (RV) is the most important cause of acute gastroenteritis (GE) requiring hospitalization of infants and young children in developed and developing countries and can be a frequent cause of death in children less than 5 years of age. GSK Biologicals has developed a vaccine against human rotavirus gastroenteritis. In this study, the immunogenicity, reactogenicity and safety of the HRV vaccine will be evaluated when stored or reconstituted in circumstances different from the recommendations: i.e. when not reconstituted with a buffer or when stored for 7 days at 37°C before reconstitution. In addition, the effect of feeding will be explored for HRV vaccine reconstituted without buffer.

DETAILED DESCRIPTION:
Assess the effect on immunogenicity of administration of vaccine without buffering agent & assess heat stability in terms of immunogenicity, reactogenicity & safety of GSK Biologicals' oral live attenuated human rotavirus (HRV) vaccine following a 0,2 m schedule, in healthy infants previously uninfected with human rotavirus

ELIGIBILITY:
INCLUSION CRITERIA:

* A male or female between, and including, 6 and 12 weeks (42-90 days) of age at the time of the first vaccination.
* Written informed consent obtained from the parent or guardian of the subject.
* Free of obvious health problems as established by medical history and clinical examination before entering into the study.

EXCLUSION CRITERIA:

* Use of any investigational or non-registered product (drug or vaccine) other than the study vaccine(s) within 30 days preceding the first dose of study vaccine or placebo, or planned use during the study period.
* Chronic administration (defined as more than 14 days) of immunosuppressants or other immune-modifying drugs prior to the first vaccine dose, since birth. (For corticosteroids, this will mean prednisone, or equivalent, greater than or equal to 0.5 mg/kg/day. Inhaled and topical steroids are allowed.)
* Planned administration of a vaccine (except routine paediatric vaccines) not foreseen by the study protocol. (If exceptionally OPV is given, this should be administered at least 14 days apart from the HRV vaccine or placebo dose.)
* Any clinically significant history of chronic gastrointestinal disease including any uncorrected congenital malformation of the GI tract or other serious medical condition as determined by the investigator.
* History of allergic disease or reactions likely to be exacerbated by any component of the vaccine.
* Any confirmed or suspected immunosuppressive or immunodeficient condition based on medical history and physical examination (no laboratory testing is required).
* Major congenital defects or serious chronic illness.
* Gastroenteritis within 7 days preceding the study vaccine administration (warrants deferral of the vaccination).
* Administration of immunoglobulins and/or blood products since birth or planned administration during the study period. Oral intake of immunoglobulins via e.g. breastfeeding is allowed.
* Previous confirmed occurrence of RV gastroenteritis.

Ages: 6 Weeks to 12 Weeks | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 450 (Actual)
Dates: Start 2005-03; Primary Completion 2005-12 (Actual); Study Completion 2005-12 (Actual)

PRIMARY OUTCOMES:
Percentage of subjects with vaccine take | At 2 months post-Dose 2

SECONDARY OUTCOMES:
Percentage of subjects who seroconverted (percentage of subjects with concentrations ≥ 20 U/mL in subjects who were negative for rotavirus (RV) before vaccination) | At 2 months post-Dose 2
Evaluation of the serum anti-RV IgA (immunoglobulin A) antibody concentrations expressed as Geometric Mean Concentrations (GMC) | At 2 months post-Dose 2
Rotavirus antigen shedding in planned stool samples | At Day 0, Day 7 and Day 15 post each study vaccine dose
Presence of RV in gastroenteritis (GE) episode stools collected | From Dose 1 of HRV vaccine/placebo up to 2 months post-Dose 2
For each type of solicited symptoms, occurrence of the symptom | Within the 15-day (Day 0-14) solicited follow-up period after each study vaccine dose
Occurrence of any Grade 2 or Grade 3 fever, vomiting or diarrhea | Within the 15-day (Day 0-14) solicited follow-up period after each study vaccine dose
Occurrence of unsolicited adverse events (AEs) according to Medical Dictionary for Regulatory Activities (MedDRA) classification | Within 31 days (Day 0-30) after each study vaccine dose
Occurrence of serious adverse events (SAEs) according to MedDRA classification | Throughout the study period (Day 0 to Month 4)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Bangkok, Thailand

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- [Background] Chokephaibulkit K et al. Immunogenicity And Vaccine Take Of RIX4414 (Rotarix") After Heat Exposure. Abstract presented at the 5th World Congress of the World Society for Pediatric infectious Diseases (WSPID). Bangkok, Thailand, 15-18 November 2007.
- [Background] Debrus S et al. Study of the viral activity of RIX4414 - human rotavirus vaccine. Abstract presented at the 47th Interscience Conference on Antimicrobial Agents and Chemotherapy (ICAAC). Chicago, USA, 17-20 September 2007.
- [Background] Debrus S et al. Viral shedding (methodology). Abstract presented at the 47th Interscience Conference on Antimicrobial Agents and Chemotherapy (ICAAC). Chicago, USA, 17-20 September 2007.
- [Background] Kerdpanich A, Chokephaibulkit K, Watanaveeradej V, Vanprapar N, Simasathien S, Phavichitr N, Bock HL, Damaso S, Hutagalung Y, Han HH. Immunogenicity of a live-attenuated human rotavirus RIX4414 vaccine with or without buffering agent. Hum Vaccin. 2010 Mar 26;6(3):10428. doi: 10.4161/hv.6.3.10428. Epub 2010 Mar 26. PMID 20220306
- [Background] Kerdpanich A et al. Feeding does not influence the immunogenicity of RIX4414 (Rotarix") in Thailand. Abstract presented at the 5th World Congress of the World Society for Pediatric infectious Diseases ( WSPID). Bangkok, Thailand, 15-18 November 2007.
- [Background] Kerdpanich et al. Exposure to elevated temperature of 37°C for 7 days does not affect immunogenicity and reactogenicity of RIX4414. Abstract presented at the 9th dsRNA Virus Meeting. Cape Town, South Africa, 21-26 October 2006.
- [Derived] Kerdpanich A, Chokephaibulkit K, Watanaveeradej V, Vanprapar N, Simasathien S, Phavichitr N, Bock HL, Damaso S, Hutagalung Y, Han HH. Immunogenicity of a human rotavirus vaccine (RIX4414) after storage at 37 degrees C for seven days. Hum Vaccin. 2011 Jan 1;7(1):74-80. doi: 10.4161/hv.7.1.13412. Epub 2011 Jan 1. PMID 21228629
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Dataset Specification: 103477 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: 103477 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: 103477 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: 103477 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: 103477 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: 103477 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register